CLINICAL TRIAL: NCT03404869
Title: Study of ORL-1M (D-mannose) in Patients With CDG-Ib
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orpha Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMID-1
Record Dates: First submitted 2018-01-13; First posted 2018-01-19 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: CDG Ib
Keywords: CDGIb MANNOSEPHOSPHATE ISOMERASE DEFICIENCY MPI DEFICIENCY PROTEIN-LOSING ENTEROPATHY-HEPATIC FIBROSIS SYNDROME SAGUENAY-LAC SAINT-JEAN SYNDROME SLSJ SYNDROME
MeSH Terms: conditions — Congenital disorder of glycosylation type 1B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (1):
- Treatment with ORL-1M - D-mannose (Other)
  Interventions: Drug: ORL-1M - D-mannose

INTERVENTIONS:
Drug: ORL-1M - D-mannose — Oral ORL-1M

SUMMARY:
Study of ORL-1M in Patients With CDG-Ib

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CGD-1b.
* Less than 18 years old.

Exclusion Criteria:

* Diagnosis of any other disease that is not a manifestation of CGD-1b.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-03-31 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in hypoglycemia, diarrhea and vomiting. | 6 months after treatment started
  Decreased frequency of hypoglycemic episode, diarrhea and vomiting frequency.

SECONDARY OUTCOMES:
Improved glycosylation pattern of serum transferrin. | 30 days after treatment started
  Normalized isoelectric focusing pattern of serum transferrin.

CONTACTS AND LOCATIONS:
Locations (1):
- Orpha Labs, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rebelo AL, Chevalier MT, Russo L, Pandit A. Role and therapeutic implications of protein glycosylation in neuroinflammation. Trends Mol Med. 2022 Apr;28(4):270-289. doi: 10.1016/j.molmed.2022.01.004. Epub 2022 Feb 1. PMID 35120836